CLINICAL TRIAL: NCT00739882
Title: A Phase IV Multicentre, Randomised, Double-blind, Placebo Controlled, Trial to Evaluate the Safety and Efficacy of Raptiva ® in the Treatment of Subjects With Moderate to Severe Plaque Psoriasis Involving Hands and/or Feet, With or Without Pustules.
Brief Title: TRUST Study: Raptiva ® in Hand & Foot Psoriasis
Acronym: TRUST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated after the European Medicines Agency recommended to suspend the marketing authorisation of Raptiva in the European Union
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 27808
Record Dates: First submitted 2008-08-20; First posted 2008-08-22 (Estimated); Results first posted 2010-08-30 (Estimated); Last update posted 2014-02-27 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Plaque Psoriasis
Keywords: Efalizumab,; Chronic plaque psoriasis; moderate to severe; involving; hands; feet
MeSH Terms: conditions — Margins of Excision

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Efalizumab (Active Comparator)
  Interventions: Drug: Efalizumab - anti CD11a recombinant human monoclonal antibody
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Efalizumab - anti CD11a recombinant human monoclonal antibody — Each subject will receive an initial conditioning dose of 0.7 mg/kg/week and then will continue treatment at a dose of 1.0 mg/kg/week. The treatment period will be 24 weeks divided into two phases: 1) double-blind for 12 weeks, and 2) open-label for 12 additional weeks, in which all subjects from the placebo group and those subjects from the Raptiva ® group with ≥ 50% of improvement will be allocated to extended treatment with Raptiva ® for 12 additional weeks while non-responders to Raptiva ® (improvement ≤ 50%) will be followed in an observational manner for 12 additional weeks without treatment.
  Arms: Efalizumab
Drug: Placebo — Placebo will be administered at Study Day (SD) 1, Week (W) 1, W 4, W 8 and W 12. Each subject will receive an initial conditioning dose of 0.7 mg/kg/week and then will continue treatment at a dose of 1.0 mg/kg/week for 12 weeks (double-blind phase)
  Arms: Placebo

SUMMARY:
To evaluate the safety and efficacy of Raptiva ® compared with placebo to control chronic moderate to severe plaque psoriasis involving the hands and/or feet scoring Physician's Global Assessment (PGA - H&F) greater-than or equal to 3 in subjects not suitable for other systemic therapies including cyclosporine, methotrexate, and Psoralen-Ultraviolet Light A (PUVA).

ELIGIBILITY:
Inclusion Criteria:

1. Subject with chronic (disease history of at least 6 months from diagnosis) moderate to severe plaque psoriasis involving the hands and/or feet (PGA - H&F ratings of 3 or 4) at screening, who have failed to respond to, or who have a contraindication to, or are intolerant to other systemic therapies including cyclosporin, methotrexate and PUVA. Subjects will be outpatients.
2. Stable disease at study entry (i.e. no exacerbation of psoriasis during the screening period).
3. At least 18 years old.
4. For women of childbearing potential, use of an acceptable method of contraception to prevent pregnancy and agreement to continue to practice an acceptable method of contraception for the duration of their participation in the study. For men, during the participation, it is mandatory to practice birth control, as there are not existing data on the effect of Raptiva ® on spermatogenesis.
5. Discontinuation of any systemic psoriasis treatment at study entry. No washout period is required for these traditional systemic psoriasis agents prior to starting study treatment.
6. Discontinuation of all biological agents at least 3 months prior to first study injection.
7. Discontinuation of any investigational drug or treatment at least 3 months prior to SD 1 or as per washout requirements from previous protocol.
8. Willingness and ability to comply with the protocol requirements for the duration of the study.
9. Written informed consent, given prior to any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw his/her consent at any time without prejudice to future medical care.

Exclusion Criteria:

1. Hypersensitivity to efalizumab or to any of the excipients
2. Current use of any prohibited therapy (systemic or topical treatments for psoriasis, immunosuppressive drugs, any other experimental drug, etc)
3. Previous or current exposure to Raptiva®
4. History of or ongoing alcohol or drug abuse
5. History of or an ongoing opportunistic infection (e.g. systemic fungal infection, parasites) or any other serious infection. This includes diagnoses that required more than 2 weeks of therapy, such as endocarditis and osteomyelitis, that have been treated in the past 6 months. In addition, if the subject is currently receiving antibiotics, antivirals, or antifungals for an infection or for suppression or prophylaxis for any diagnosis, the subject will be excluded.
6. Seropositivity for hepatitis B antigen, hepatitis C antibody, or human immunodeficiency virus (HIV). Subjects will undergo testing during screening, and any subjects who are seropositive for hepatitis B antigen, hepatitis C antibody, or HIV will be excluded.
7. History of active or latent tuberculosis within one year prior to screening (to be determined by assessment according to national and/or local recommendation).
8. Presence or history of malignancy, including lymphoproliferative disorders.
9. Pregnancy or breast-feeding
10. History of hepatic cirrhosis, regardless of cause or severity
11. History of thrombocytopenia, haemolytic anaemia, clinically significant anaemia, a white blood cell count <4,000 cells/μL or >14,000 cells/μL, a haematocrit (HCT) <30% or a haemoglobin (Hgb) level <11 g/dL, a platelet count <150,000 cells/μL
12. Hepatic enzyme levels ≥3 times the upper limit of normal or serum creatinine level ≥2 times the upper limit of normal
13. Vaccination with a live or live-attenuated virus or live or live-attenuated bacteria vaccine within the 14 days prior to the first dose of Raptiva®
14. Any medical condition that, in the judgment of the Investigator, would jeopardise the subject's safety following exposure to investigational medicinal product (Raptiva® or placebo equivalent) or would significantly interfere with the Subject's ability to comply with the provisions of this protocol.
15. Other specific forms of psoriasis like guttate, erythrodermic or pustular psoriasis as sole or predominant for of psoriasis.
16. Immunodeficiencies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Selenko-Gebauer, MD, Study Director — Merck Serono S.A., Geneva
Locations (1):
- University of Vienna Medical School, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject's first visit: 08 April 2008, last subject's last visit: 15 June 2009. Seventy six subjects entered the study, 46 completed the double-blind period and 31 of these then entered the open-label period. The remaining 15 entered an observational follow-up.
Pre-assignment Details: During the screening period, approximately 200 subjects were to be screened for trial eligibility within 14 days before Day 1. A total of 100 subjects had been screened at the time the trial was terminated, of whom 76 subjects were enrolled in the trial.
Groups:
- Efalizumab: Each subject will receive an initial conditioning dose of 0.7 mg/kg/week and then will continue treatment at a dose of 1.0 mg/kg/week. The treatment period will be 24 weeks divided into two phases: 1) double-blind for 12 weeks, and 2) open-label for 12 additional weeks, in which all subjects from the placebo group and those subjects from the Raptiva ® group with ≥ 50% of improvement will be allocated to extended treatment with Raptiva ® for 12 additional weeks while non-responders to Raptiva ® (improvement ≤ 50%) will be followed in an observational manner for 12 additional weeks without treatment.
Period: Double-blind Period
Arm/Group | Efalizumab | Placebo
Started | 51 | 25
Completed | 32 | 14
Not Completed | 19 | 11
Not completed — Adverse Event | 1 | 2
Not completed — Protocol Violation | 1 | 0
Not completed — Lack of Efficacy | 1 | 1
Not completed — Other | 16 | 8
Period: Open-label Period
Arm/Group | Efalizumab | Placebo
Started | 17 | 14
Completed | 7 | 9
Not Completed | 10 | 5
Not completed — Adverse Event | 1 | 0
Not completed — Other | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efalizumab | Placebo | Total
Number analyzed (Participants) | 51 | 25 | 76
Age, Customized [Number; unit: participants]
  18-40 years | 16 | 4 | 20
  41-64 years | 29 | 17 | 46
  >64 years | 6 | 4 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (13.3) | 51.7 (12.9) | 49.9 (13.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 10 | 31
  Male | 30 | 15 | 45
Region of Enrollment [Number; unit: participants]
  Austria | 7 | 4 | 11
  Belgium | 4 | 0 | 4
  France | 8 | 5 | 13
  Germany | 14 | 4 | 18
  Italy | 2 | 2 | 4
  Netherlands | 0 | 2 | 2
  Spain | 7 | 4 | 11
  Turkey | 9 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Proportion Of Participants Achieving A Physician's Global Assessment - Hand & Foot (PGA - H&F) Rating Of Clear, Almost Clear Or Mild At Week 12
Description: The proportion of subjects achieving a PGA - H&F rating of clear, almost clear, or mild at Week 12:
  Clear - No signs of plaque psoriasis on the hands and/or feet; Almost Clear - Just perceptible erythema and just perceptible scaling on the hands and/or feet; Mild - Light pink erythema with minimal scaling and with or without pustules on the hands and/or feet
Time Frame: 12 weeks
Population: Due to the termination of the trial, analysis of efficacy-related endpoints was not performed
Arm/Group | Efalizumab | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Proportion Of Participants Achieving A Physician's Global Assessment - Hand & Foot (PGA - H&F) Rating Of Clear, Or Almost Clear At Week 12
Description: The proportion of participants achieving a PGA - H&F rating of clear, or almost clear, at Week 12:
  Clear - No signs of plaque psoriasis on the hands and/or feet; Almost Clear - Just perceptible erythema and just perceptible scaling on the hands and/or feet
Time Frame: 12 weeks
Population: Due to the termination of the trial, analysis of efficacy-related endpoints was not performed
Arm/Group | Efalizumab | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Proportion Of Participants Achieving A Physician's Global Assessment - Hand & Foot (PGA - H&F) Rating Of Clear, Almost Clear Or Mild At Week 24
Description: The proportion of participants achieving a PGA - H&F rating of clear, almost clear, or mild at Week 24:
  Clear - No signs of plaque psoriasis on the hands and/or feet; Almost Clear - Just perceptible erythema and just perceptible scaling on the hands and/or feet; Mild - Light pink erythema with minimal scaling and with or without pustules on the hands and/or feet
Time Frame: 24 weeks
Population: Due to the termination of the trial, analysis of efficacy-related endpoints was not performed
Arm/Group | Efalizumab | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Proportion of Participants From the Initial Placebo Group Achieving a PGA - H&F of Rating of Clear, Almost Clear, or Mild From Week 12 to Week 24.
Description: The proportion of participants achieving a PGA - H&F rating of clear, or almost clear, at Week 24:
  Clear - No signs of plaque psoriasis on the hands and/or feet; Almost Clear - Just perceptible erythema and just perceptible scaling on the hands and/or feet; Mild - Light pink erythema with minimal scaling and with or without pustules on the hands and/or feet
Time Frame: 24 weeks
Population: Due to the termination of the trial, analysis of efficacy-related endpoints was not performed
Arm/Group | Efalizumab | Placebo
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Proportion Of Participants Achieving A Physician's Global Assessment (PGA) Rating of Good, Excellent, Or Cleared At Week 12
Description: The proportion of participants achieving a PGA rating of good, excellent, or cleared at Week 12.
  Cleared = 100% improvement; Excellent = 75-99% improvement; Good = 50-74% improvement
Time Frame: 12 weeks
Population: Due to the termination of the trial, analysis of efficacy-related endpoints was not performed
Arm/Group | Efalizumab | Placebo
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Proportion Of Participants Achieving A Physician's Global Assessment (PGA) Rating of Excellent, Or Cleared At Week 12
Description: The proportion of participants achieving a PGA rating of excellent, or cleared at Week 12.
  Cleared = 100% improvement; Excellent = 75-99% improvement
Time Frame: 12 weeks
Population: Due to the termination of the trial, analysis of efficacy-related endpoints was not performed
Arm/Group | Efalizumab | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events occurring during the 12-week double-blind period and the 12-week open-label period are reported
Description: Treatment-emergent adverse events are reported. 'Other Adverse Events' table shows the number of participants experiencing any adverse event and the listing shows all adverse events occurring above the reporting threshold during the double-blind period and open-label period.
Arm/Group | Efalizumab - Double-blind Period | Placebo - Double-blind Period | Efalizumab - Open-label Period | Placebo - Open-label Period
Serious Adverse Events (participants affected / at risk) | 1/51 | 1/25 | 0/17 | 2/14
Other Adverse Events (participants affected / at risk) | 35/51 | 13/25 | 8/17 | 7/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab - Double-blind Period (N=51) | Placebo - Double-blind Period (N=25) | Efalizumab - Open-label Period (N=17) | Placebo - Open-label Period (N=14)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Tendon operation (Surgical and medical procedures) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efalizumab - Double-blind Period (N=51) | Placebo - Double-blind Period (N=25) | Efalizumab - Open-label Period (N=17) | Placebo - Open-label Period (N=14)
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Acute tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Conjunctival hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1
Eye swelling (Eye disorders) | 1 | 0 | 0 | 0
Eyelid oedema (Eye disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 5 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal infection (Infections and infestations) | 2 | 0 | 0 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 10 | 1 | 1 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 2 | 0 | 0 | 0
Influenza like illness (General disorders) | 5 | 1 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 6 | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Meningitis aseptic (Infections and infestations) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 3 | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 2 | 0 | 0
Oral mucosa erosion (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 1 | 0 | 0 | 0
Sinus congestion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tendon operation (Surgical and medical procedures) | 0 | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
Following the recommendation of the European Medicines Agency (EMEA) to suspend the marketing authorization of Raptiva® and the subsequent premature termination of this trial analysis of efficacy-related endpoints was not performed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other